CLINICAL TRIAL: NCT05899764
Title: Epileptic Hippocampus in Alzheimer's Disease
Acronym: EHAD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Keith Vossel, Center Director at the Mary S. Easton Center for Alzheimer's Disease Research and Professor of Neurology, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-001000
Record Dates: First submitted 2023-03-21; First posted 2023-06-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Alzheimer's Disease; Mild Cognitive Impairment; Epileptic Activity; Pathological High Frequency Oscillations; Depth Electrode; Brivaracetam
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BRIV Experimental (Experimental): 25 subjects with MCI or AD who meet inclusion criteria will receive the drug: brivaracetam. A scalp EEG will record their brain activity for 6 days at the hospital. On nights 4 and 5, we will intravenously administer brivaracetam. Doses will vary depending on their effects on epileptic activity. We will determine whether brivaracetam 25 mg IV suppresses the number of epileptic events and pHFOs by >50%, which is analogous to our preclinical investigations with this drug in AD models. If the 50% suppression is reached, the same dosage will be repeated the following night to ensure reproducibility. If the 50% suppression is not reached, then the dosage of brivaracetam will be increased to 50 mg the following night. Once the depth electrode is surgically removed, subjects will go home with a supply of brivaracetam. They will take the drug for 12 months.
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — * Intravenous administration: 25 mg or 50 mg will be administered depending on its effects on epileptic activity during a hospital stay where simultaneous EEG and depth electrode recordings will be measuring epileptic activity.
  * Oral administration: Subjects will take 25mg or 50mg twice a day for 12 months. The dosage will depend on its effects on epileptic activity. Brivaracetam levels will be measured on months 3, 6 and 12.
  Other Names: Briviact; Brivajoy

SUMMARY:
The major goals of the study are to 1) characterize hippocampal activity in patients with mild cognitive impairment (MCI) due to Alzheimer's disease (AD) and AD who have suspected hippocampal epileptic activity based on scalp EEG recordings from IRB # 21-001603; 2) study the efficacy of brivaracetam to suppress epileptic activity and pathological high frequency oscilations (pHFOs) during hippocampal depth electrode and scalp EEG in patients with MCI and AD; and 3) investigate the effects of brivaracetam on cognition in an open-label pilot study.

DETAILED DESCRIPTION:
This is a prospective, single-center, open-label, pilot study. Individuals with mild cognitive impairment (MCI) and Alzheimer's disease (AD) who show epileptic activity as part of an overnight EEG from study IRB#21-001603 or as a part of a clinical EEG will be eligible. After informed consent, participants will undergo hippocampal depth electrode placement and full scalp electroencephalogram (EEG) recordings to characterize epileptic hippocampal activity and pathological high frequency oscilations (pHFOs). During recordings, the investigators will determine whether brivaracetam, given intravenously, suppresses epileptic activity/high frequency oscillations. After recordings are completed, investigators will test whether brivaracetam, in oral tablets, improves cognition over the course of 1 year. Participants will include men and women 45-70 years of age who meet criteria for MCI due to AD and mild AD. Clinical diagnoses will be made by a panel of experts. The target enrollment for the 5-year period is 25 participants. The ratio of males to females is nearly equal, given previous experience of the investigators in finding subclinical epileptiform activity in both males and females with AD. The findings may lead to better characterization of neural network dysfunction in Alzheimer's disease and identify subpopulations with subclinical epileptiform activity or seizures and cognitive impairments who could benefit from antiseizure therapies. This study also has the potential of advancing our knowledge of the pathophysiology of Alzheimer's disease.

If epileptic activity or pHFOs are identified during an overnight EEG from study Biomarkers in Neurodegenerative Disease (UCLA IRB#21-001603) or through a clinical study, the investigators will offer the opportunity to be part of this research study. Consenting and study overview will be conducted by the investigators. If accepted into the study, participants will undergo a magnetic resonance venography (MRV), magnetic resonance angiography (MRA) and a gadolinium-enhanced MRI a couple of weeks prior the hippocampal implantation of one or two depth electrodes. A coagulation blood draw will be collected prior to the surgery during one of the neuroimaging visits. Before the surgical procedure, participants will complete cognitive testing with one of the investigators. The Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog), Stroop Interference naming, and Virtual Route Learning Test (VRLT) will be collected. If coagulation levels come back normal and the participants are in good health, they will undergo general anesthesia and a neurosurgeon will implant one to two depth electrodes in the hippocampus. A Leksell stereotactic frame will be attached to the head to guide localization and a CT angiography will be collected to guide the surgical procedure. Participants will go to the Intensive Care Unit and spend the night there while their recovery is being monitored.

The next day, a scalp EEG will be placed to record brain activity for six days and five nights in conjunction with the hippocampal depth electrode(s) already implanted. On nights four and five, participants will undergo intravenous administration of brivaracetam to study its effects on hippocampal epileptic activity. Investigators will determine whether brivaracetam 25 mg IV suppresses the number of epileptic events and pHFOs by >50%, which is analogous to preclinical investigations with this drug in AD models. If the 50% suppression is reached, the same dosage will be repeated the following night to ensure reproducibility. If the 50% suppression is not reached, then the dosage of brivaracetam will be increased to 50 mg the following night. On day six, the depth electrode will be removed using local anesthesia. Participants will stay at the hospital one more day for recovery and will be discharged on day seven.

Participants will take brivaracetam twice a day for 1 year and will come back the University of California, Los Angeles (UCLA) at 3 months, 6 months, and 1 year to complete cognitive testing (ADAS-cog, Stroop Interference naming, and VRLT) and receive additional brivaracetam supplies. During the follow-up visits, blood samples will be collected to study plasma biomarkers of neurodegenerative diseases. Participants will conclude their participation after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Meet research criteria for mild cognitive impairment (Albert et al. 2011) or Alzheimer's disease (McKhann et al. 2011) with high biomarker probability of Alzheimer's disease pathophysiology
* Ages 45 to 70
* Epileptic activity and/or pHFOs in temporal or fronto-temporal electrodes
* Willing and able informant who has at least weekly contact with subject
* Mini-Mental State Examination score of 18 or greater and/or Clinical Dementia Rating less than 2. These two examinations will be obtained from their participation in UCLA IRB#21-001603 or will be collected if subjects are referred by a clinician.

Exclusion Criteria:

1. Risk factors for epileptic activity besides neurodegenerative disease
2. Concurrent use of antiseizure medications
3. Severe periventricular white matter disease
4. Clinically significant lacunar infarcts
5. Anticoagulant use
6. Significant systemic medical illness:

   * History of Korsakoff's syndrome
   * Alcohol or substance abuse preceding dementia & still present within 5 years of onset
   * Untreated vitamin B12 or folate deficiency
   * History of head trauma with persistent deficits
   * Untreated syphilis
   * History of multiple sclerosis or another neuro-inflammatory disorder
   * History of vascular or multi-infarct dementia
   * Diagnosis of Huntington's disease
   * History of normal pressure hydrocephalus
   * History of CNS lesions deemed to be clinically significant
   * Unresolved or present subdural hematoma
   * History of intracerebral hemorrhage
   * Systematic liver disease
   * Renal insufficiency requiring dialysis
   * Encephalitis or meningitis
   * Severe white matter disease as defined by a score of 3 on the age-related white matter changes scale
   * Lacunar infarcts deemed to be clinically significant
   * Cortical stroke
   * Respiratory condition requiring oxygen
   * Untreated hypothyroidism
7. Any other medical condition which is determined by the investigators to potentially create an undue risk for an adverse event
8. Use of medications likely to affect CNS functions (e.g., benzodiazepines, narcotics). Patients are allowed to take cholinesterase inhibitors and memantine as long as the dosage is stable for 30 days prior to study entry.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Brivaracetam on Cognition | 3 months
  To determine the efficacy of brivaracetam to improve cognitive function for the following task at 3 months while taking brivaracetam oral tablets: Stroop interference naming (number correct)
Brivaracetam on Cognition | 3 months
  To determine the efficacy of brivaracetam to improve cognitive function for the following task at 3 months while taking brivaracetam oral tablets: Virtual Route Learning Test (VRLT)

SECONDARY OUTCOMES:
Brivaracetam on Cognition | 12 months
  To determine the efficacy of brivaracetam to improve cognitive function in the following task while taking brivaracetam oral tablets: Stroop interference naming (number correct) at 6 and 12 months
Brivaracetam on Cognition | 12 months
  To determine the efficacy of brivaracetam to improve cognitive function in the following task while taking brivaracetam oral tablets: Virtual Route Learning Test at 6 and 12 months
Brivaracetam on Cognition | 12 months
  To determine the efficacy of brivaracetam to improve cognitive function in the following task while taking brivaracetam oral tablets: Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) at 3, 6, and 12 months (12 month data will be compared to historical data from MCI and AD participants in the Alzheimer's Disease Neuroimaging Initiative)
Brivaracetam on Functional Decline | 12 months
  To compare the rate of decline measured by clinical dementia rating - sum of boxes (CDR-SB) at 12 months while taking brivaracetam to the historical rate of decline in MCI and AD participants collected through the Alzheimer's Disease Neuroimaging Initiative
Brivaracetam and Plasma Biomarkers | 12 months
  To determine whether brivaracetam improves levels of plasma biomarkers of neurodegenerative diseases: Abeta 42/Abeta 40 at 3 months, 6 months, and 12 months while participants take brivaracetam
Brivaracetam and Plasma Biomarkers | 12 months
  To determine whether brivaracetam improves levels of plasma biomarkers of neurodegenerative diseases: total tau at 3 months, 6 months, and 12 month while participants take brivaracetam
Brivaracetam and Plasma Biomarkers | 12 months
  To determine whether brivaracetam improves levels of plasma biomarkers of neurodegenerative diseases: p-tau at 3 months, 6 months, and 12 month while participants take brivaracetam
Brivaracetam and Plasma Biomarkers | 12 months
  To determine whether brivaracetam improves levels of plasma biomarkers of neurodegenerative diseases: GFAP at 3 months, 6 months, and 12 month while participants take brivaracetam
Brivaracetam and Plasma Biomarkers | 12 months
  To determine whether brivaracetam improves levels of plasma biomarkers of neurodegenerative diseases: NfL at 3 months, 6 months, and 12 month while participants take brivaracetam

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Vossel, MD, MSc, Principal Investigator — Mary S. Easton Center at UCLA
Locations (1):
- Mary S. Easton Center for Alzheimer's Research and Care, Los Angeles, California, United States

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Stephen LJ, Brodie MJ. Brivaracetam: a novel antiepileptic drug for focal-onset seizures. Ther Adv Neurol Disord. 2017 Nov 23;11:1756285617742081. doi: 10.1177/1756285617742081. eCollection 2018. PMID 29399049
- [Background] Vossel KA, Beagle AJ, Rabinovici GD, Shu H, Lee SE, Naasan G, Hegde M, Cornes SB, Henry ML, Nelson AB, Seeley WW, Geschwind MD, Gorno-Tempini ML, Shih T, Kirsch HE, Garcia PA, Miller BL, Mucke L. Seizures and epileptiform activity in the early stages of Alzheimer disease. JAMA Neurol. 2013 Sep 1;70(9):1158-66. doi: 10.1001/jamaneurol.2013.136. PMID 23835471
- [Background] Vossel KA, Ranasinghe KG, Beagle AJ, Mizuiri D, Honma SM, Dowling AF, Darwish SM, Van Berlo V, Barnes DE, Mantle M, Karydas AM, Coppola G, Roberson ED, Miller BL, Garcia PA, Kirsch HE, Mucke L, Nagarajan SS. Incidence and impact of subclinical epileptiform activity in Alzheimer's disease. Ann Neurol. 2016 Dec;80(6):858-870. doi: 10.1002/ana.24794. Epub 2016 Nov 7. PMID 27696483
- [Result] Vossel K, Ranasinghe KG, Beagle AJ, La A, Ah Pook K, Castro M, Mizuiri D, Honma SM, Venkateswaran N, Koestler M, Zhang W, Mucke L, Howell MJ, Possin KL, Kramer JH, Boxer AL, Miller BL, Nagarajan SS, Kirsch HE. Effect of Levetiracetam on Cognition in Patients With Alzheimer Disease With and Without Epileptiform Activity: A Randomized Clinical Trial. JAMA Neurol. 2021 Nov 1;78(11):1345-1354. doi: 10.1001/jamaneurol.2021.3310. PMID 34570177